CLINICAL TRIAL: NCT06339073
Title: CT-based Model for Predicting Prolonged Weaning From Mechanical Ventilation in Patients With Abdominal Trauma: a Retrospective Cohort Study
Brief Title: CT-based Model for Predicting Prolonged Weaning in Patients With Abdominal Trauma
Status: Completed | Type: Observational
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Fengchan Xi, Chief of the Department of Intensive Care Unit, Associate chiefphysician, Nanjing Maternity and Child Health Care Hospital
Other Study IDs: 2021NZKY-045-01
Record Dates: First submitted 2024-03-24; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Wounds and Injuries; Ventilation Therapy; Complications
Keywords: computed tomography; prolonged weaning; ventilation; trauma
MeSH Terms: conditions — Wounds and Injuries; Respiratory Aspiration | interventions — Respiration, Artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: mechanical ventilation — Abdominal trauma patients were treated with mechanical ventilation according to their conditions.

SUMMARY:
Critically ill patients often require tracheal intubation for mechanical ventilation, and timely weaning is crucial for airway management and reducing complications. However, there is currently a lack of an effective tool to predict weaning time in critically ill patients. This retrospective study established an effective nomogram model for predicting the time of weaning from mechanical ventilation in abdominal trauma patients by considering multiple perspectives. The model has been validated and demonstrated good performance in terms of discrimination, calibration, and clinical utility. Moreover, the model can effectively predict the prognosis of critically ill patients. The findings of this study have important implications for guiding respiratory management in clinically critically ill patients, particularly trauma patients.

ELIGIBILITY:
Inclusion Criteria:

* (1) with information on survival status and time;
* (2) aged 18-80 years;
* (3) admitted to ICU;
* (4) with abdominal CT performed within 1-week post-trauma;
* (5) use of mechanical ventilation.

Exclusion Criteria:

* (1) low-quality CT images;
* (2) history of mental illness.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with abdominal trauma admitted to the General Surgical Department of Jinling Hospital from January 2010 to April 2023 were screened for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 1023 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Prolonged mechanical ventilation | through whole hospitalization of each participant, an average of 25 days
  Prolonged mechanical ventilation was defined as length of mechanical ventilation >7 days

CONTACTS AND LOCATIONS:
Locations (1):
- the General Surgical Department of Jinling Hospital, Nanjing, Jiangsu, China